CLINICAL TRIAL: NCT05255458
Title: A Phase 3 Clinical Study Evaluating the Long-term Efficacy and Safety of AK102 in Patients With Primary Hypercholesterolemia and Mixed Hyperlipidemia
Brief Title: A Study to Evaluate the Long-term Efficacy and Safety of AK102 in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK102-303
Record Dates: First submitted 2022-02-09; First posted 2022-02-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK102 regimen 1 (Experimental)
  Interventions: Biological: AK102
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AK102 — Administered AK102 by subcutaneous injection Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: AK102 regimen 1
Drug: Placebo — Administered placebo by subcutaneous injection Drug: Statins and/or Ezetimibe lipid-lowering therapies
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase 3 clinical study evaluating the long-term efficacy and safety of AK102 in patients with primary hypercholesterolemia and mixed hyperlipidemia.

DETAILED DESCRIPTION:
This is a Phase 3 clinical study to evaluate the long-term efficacy and safety of AK102, a monoclonal antibody, against proprotein convertase subtilisin/kexin type 9 (PCSK9), in subjects with primary hypercholesterolemia and mixed hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject understand and voluntarily sign the written Inform Consent Form (ICF), which must be signed before performing the study procedures.
2. Male or female patients aged between 18 and 80 years (including upper and lower limits).
3. The fasting serum LDL-C level of subjects did not meet the treatment goal after at least 4 weeks of stable lipid-lowering background treatment.
4. Triglyceride ≤ 4.5 mmol/L (400 mg/dl).

Exclusion Criteria:

1. Homozygous Familial Hypercholesterolemia (HoFH).
2. Received PCSK9 inhibitors within 6 months before randomization.
3. Known sensitivity to PCSK9 inhibitors and any substances to be administered.
4. Severe liver and renal dysfunction.
5. Previously received organ transplantation.
6. Uncontrolled hypothyroidism or hyperthyroidism.
7. Uncontrolled hypertension.
8. Known hyperlipidemia secondary to comorbidity, including nephrotic syndrome, cholestatic liver failure, etc.
9. History of malignancy of any organ system within the past 5 years.
10. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Precentage change from baseline of serum LDL-C level | At week 52
The incidence and severity of adverse events (AE) | Week 0-52

SECONDARY OUTCOMES:
Value and percentage change from baseline of serum TC levels | Week 0-52
Value and percentage change from baseline of serum TG levels | Week 0-52
Value and percentage change from baseline of serum non HDL-C levels | Week 0-52
Value and percentage change from baseline of serum ApoB levels | Week 0-52
Value and percentage change from baseline of serum HDL-C levels | Week 0-52
Value and percentage change from baseline of serum ApoA-I levels | Week 0-52
Value and percentage change from baseline of serum Lp(a) levels | Week 0-52
Evaluate the population pharmacokinetic (PK) characteristics of AK102 , such as AK102 concentration | Week 0-52
Number and percentage of subjects with positive anti-AK102 antibody (ADA) / neutralizing antibody (NAB) and the time of ADA / nab positivity | Week 0-52

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Hospital of Nanchang, Nanchang, Jiangxi, China